CLINICAL TRIAL: NCT00972517
Title: Safety and Immunogenicity Study of GSK Biologicals' Pandemic Influenza Candidate Vaccine (GSK2340272A) in Children Aged 3 to 17 Years
Brief Title: Study to Evaluate the Immunogenicity and Safety of an Investigational Influenza Vaccine (H1N1) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 113638; 2009-015011-41 (EudraCT Number)
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340272A; influenza infection
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- Group A (Experimental): Subjects receiving alternative dose of GSK23440272A vaccine
  Interventions: Biological: GSK investigational vaccine GSK2340272A

INTERVENTIONS:
Biological: GSK investigational vaccine GSK2340272A — Three intramuscular injections

SUMMARY:
The objective of this study is to evaluate the immunogenicity and safety of GSK Biologicals' investigational vaccine GSK2340272A in children aged between 3 and 17 years.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol amendment 1, October 2009. The impacted section are the study design section, the outcomes measures section and the intervention section.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* Children, male or female, aged between 3 and 17 years at the time of the first study vaccination.
* Written informed consent obtained from the subject parent(s) or LAR(s) of the subject. Assent obtained from the subject when applicable.
* Healthy children as established by medical history and clinical examination when entering into the study.
* Parent/LAR with access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Clinically or virologically confirmed influenza infection within six months preceding the study start.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* Previous administration of any H1N1 A/California-like vaccine.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned during the study.
* If the subject is female and if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after completion of the vaccination series.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Known use of an analgesic or antipyretic medication within 12 hours prior to first vaccination.
* Child in Care.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2009-09-29 (Actual); Primary Completion 2010-11-22 (Actual); Study Completion 2010-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Germany (8):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Garcia-Sicilia J, Gillard P, Carmona A, Tejedor JC, Aristegui J, Merino JM, Behre U, Caplanusi A, Vaman T, Dieussaert I. Immunogenicity and safety of AS03-adjuvanted H1N1 pandemic vaccines in children and adolescents. Vaccine. 2011 Jun 10;29(26):4353-61. doi: 10.1016/j.vaccine.2011.04.011. Epub 2011 Apr 17. PMID 21504774
- [Background] Garcia-Sicilia J, Aristegui J, Omenaca F, Carmona A, Tejedor JC, Merino JM, Garcia-Corbeira P, Walravens K, Bambure V, Moris P, Caplanusi A, Gillard P, Dieussaert I. Safety and persistence of the humoral and cellular immune responses induced by 2 doses of an AS03-adjuvanted A(H1N1)pdm09 pandemic influenza vaccine administered to infants, children and adolescents: Two open, uncontrolled studies. Hum Vaccin Immunother. 2015;11(10):2359-69. doi: 10.1080/21645515.2015.1063754. PMID 26176592
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One subject was enrolled but not vaccinated and therefore, was not included in the number of subjects under "STARTED"
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Flu BS1_3-5 Years Group: Subjects 3 to 5 years of age, received 2 doses of the GSK2340272A vaccine (Flu) at Day 0 and Day 21 with blood sampling schedule as follows: On Day 0 (before the first vaccination); On Day 21 (before the second vaccination); On Day 42 (21 days after the second vaccination); At Month 6 (6 months after the first vaccination).
- Flu BS1_6-9 Years Group: Subjects 6 to 9 years of age, received 2 doses of the GSK2340272A vaccine (Flu) at Day 0 and Day 21 with blood sampling schedule as follows: On Day 0 (before the first vaccination); On Day 21 (before the second vaccination); On Day 42 (21 days after the second vaccination); At Month 6 (6 months after the first vaccination).
- Flu BS1_10-17 Years Group: Subjects 10 to 17 years of age, received 2 doses of the GSK2340272A vaccine (Flu) at Day 0 and Day 21 with blood sampling schedule as follows: On Day 0 (before the first vaccination); On Day 21 (before the second vaccination); On Day 42 (21 days after the second vaccination); At Month 6 (6 months after the first vaccination).
- Flu BS2_3-5 Years Group: Subjects 3 to 5 years of age, received 2 doses of the GSK2340272A vaccine (Flu) at Day 0 and Day 21 with blood sampling schedule as follows: On Day 42 (21 days after the second vaccination); At Month 6 (6 months after the first vaccination); At Month 12 (one year after the first vaccination).
- Flu BS2_6-9 Years Group: Subjects 6 to 9 years of age, received 2 doses of the GSK2340272A vaccine (Flu) at Day 0 and Day 21 with blood sampling schedule as follows: On Day 42 (21 days after the second vaccination); At Month 6 (6 months after the first vaccination); At Month 12 (one year after the first vaccination).
- Flu BS2_10-17 Years Group: Subjects 10 to 17 years of age, received 2 doses of the GSK2340272A vaccine (Flu) at Day 0 and Day 21 with blood sampling schedule as follows: On Day 42 (21 days after the second vaccination); At Month 6 (6 months after the first vaccination); At Month 12 (one year after the first vaccination).
Period: Overall Study
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Started | 31 | 31 | 60 | 30 | 34 | 58
Completed | 31 | 30 | 60 | 27 | 33 | 58
Not Completed | 0 | 1 | 0 | 3 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group A
Number analyzed (Participants) | 244
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 9.2 (4.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 128

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibody Titers Against the Flu A/California/7/2009 (H1N1) Vaccine Strain
Description: Antibody titers were expressed as Geometric mean titers (GMTs).
Time Frame: At Day 0, Day 21 and Day 42
Population: The ATP cohort for immunogenicity included all subjects for whom 2 doses were administrated and assay results were available for the blood samples taken before the first vaccination (Day 0), before the second vaccination (Day 21) and after the second vaccine dose (Day 42). No blood samples were planned at Day 0 and Day 21 for Flu BS2 Groups.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 28 | 30 | 54 | 25 | 30 | 57
Titers
  H1N1, Day 0: number analyzed (Participants) | 28 | 30 | 54 | 0 | 0 | 0
  H1N1, Day 0 | 5.7 [4.5 to 7.2] | 5.2 [4.8 to 5.8] | 9.9 [7 to 14.1] |  |  |
  H1N1, Day 21: number analyzed (Participants) | 28 | 30 | 54 | 0 | 0 | 0
  H1N1, Day 21 | 192.6 [145.6 to 254.8] | 190.3 [147 to 246.3] | 479.3 [361.8 to 634.9] |  |  |
  H1N1, Day 42 | 1361.7 [1107 to 1674.9] | 970.1 [765.8 to 1228.8] | 1069.4 [892.6 to 1281.3] | 1161.7 [905.2 to 1490.9] | 915.7 [759.1 to 1104.6] | 979.6 [845.3 to 1135.2]

2. Primary Outcome: Number of Seroconverted Subjects for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titre less than (<) 1:10 and a post-vaccination titre greater than or equal to (≥) 1:40 or a pre-vaccination titre ≥ 1:10 and at least a 4-fold increase in post-vaccination titre. The Committee for Medicinal Products for Human Use (CHMP) criterion was fulfilled if the point estimate for SCR was greater than (>) 40% in children aged 3 to 17 years.
Time Frame: At Day 42
Population: This measure was assessed on the ATP cohort for immunogenicity on subjects with assay results available for Day 0, Day 21 and Day 42. As no pre-vaccination (Day 0 and Day 21) blood samples were planned for the Flu BS2 Groups, seroconversion at Day 42 could not be computed for those groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group
Number analyzed (Participants) | 28 | 30 | 54
Participants | 28 | 30 | 53

3. Primary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titre greater than or equal to (≥) 1:40, that usually is accepted as indicating protection. The Committee for Medicinal Products for Human Use (CHMP) criterion was fulfilled if the post-vaccination time point estimate for SPR the point estimate for SPR was greater than (>) 70% in children aged 3 to 17 years.
Time Frame: At Day 42
Population: The ATP cohort for immunogenicity included all evaluable subjects for whom 2 doses were administrated and assay results were available for antibodies against H1N1 antigen for the blood sample taken after the second vaccine dose (Day 42).
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 28 | 30 | 54 | 25 | 30 | 57
Participants | 28 | 30 | 54 | 25 | 30 | 57

4. Primary Outcome: HI Antibody Geometric Mean Fold Rise (GMFR) Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: GMFR, also called seroconversion factor (SCF), was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The CHMP criterion was fulfilled if the point estimate for GMFR was greater than (>) 2.5 in children aged 3 to 17 years
Time Frame: At Day 42
Population: This measure was assessed on the ATP cohort for immunogenicity on subjects with assay results available for Day 0, Day 21 and Day 42. As no pre-vaccination (Day 0 and Day 21) blood samples were planned for the Flu BS2 Groups, GMFR at Day 42 could not be computed for those groups.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group
Number analyzed (Participants) | 28 | 30 | 54
Fold change | 237.68 [175.28 to 322.29] | 185.25 [142.09 to 241.52] | 107.74 [76.64 to 151.45]

5. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibody Titers Against the Flu A/California/7/2009 (H1N1) Vaccine Strain
Description: Antibody titers were expressed as geometric mean titers (GMTs)
Time Frame: At Month 6
Population: The ATP cohort for antibody persistence at Month 6 included all evaluable subjects for whom data concerning immunogenicity outcome measures were available for antibodies against the study vaccine antigen component at Month 6.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 27 | 28 | 53 | 23 | 27 | 47
Titers | 140.8 [118.2 to 167.6] | 154.2 [126.5 to 187.9] | 254.6 [199 to 325.7] | 129.4 [94.6 to 176.9] | 148.2 [119 to 184.4] | 243.6 [185.9 to 319.3]

6. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibody Titers Against the Flu A/California/7/2009 (H1N1) Vaccine Strain
Description: Antibody titers were expressed as geometric mean titers (GMTs)
Time Frame: At Month 12
Population: The ATP cohort for antibody persistence at Month 12 including all evaluable subjects for whom assay results were available for antibodies against the study vaccine antigen component at Month 12. As no blood samples were planned at Month 12 for the Flu BS1 Groups, GMTs could not be computed for those groups.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 20 | 26 | 41
Titers | 48.5 [35.7 to 65.7] | 60.5 [49.2 to 74.3] | 132.8 [94.9 to 185.8]

7. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 2
Time Frame: At Month 6
Population: The ATP cohort for antibody persistence at Month 6 including all evaluable subjects for whom assay results were available at pre-vaccination time points (Day 0 and Day 21) and post-vaccination time point (Month 6). No pre-vaccination blood samples were taken from Flu BS2 Groups and hence seroconversion could not be assessed for these groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group
Number analyzed (Participants) | 27 | 28 | 53
Participants | 27 | 28 | 50

8. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 3
Time Frame: At Month 6
Population: The ATP cohort for antibody persistence at Month 6 including all evaluable subjects for whom assay results were available for antibodies against the study vaccine antigen component at Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 27 | 28 | 53 | 23 | 27 | 47
Participants | 27 | 28 | 53 | 20 | 27 | 47

9. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 3
Time Frame: At Month 12
Population: The ATP cohort for antibody persistence at Month 12 including all evaluable subjects for whom assay results were available for antibodies against the study vaccine antigen component at Month 12. As no blood samples were planned at Month 12 for the Flu BS1 Groups, no data were computed for these groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 20 | 26 | 41
Participants | 17 | 22 | 37

10. Secondary Outcome: HI Antibody Geometric Mean Fold Rise (GMFR) Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 4
Time Frame: At Month 6
Population: The ATP cohort for antibody persistence at Month 6 including all subjects for whom assay results were available for antibodies against the study vaccine antigen component pre-vaccination (Day 0 and Day 21) and at Month 6. As no pre-vaccination blood samples were planned for the Flu BS2 Groups, GMFR at Month 6 could not be computed for those groups.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group
Number analyzed (Participants) | 27 | 28 | 53
Fold change | 27.44 [22.42 to 33.57] | 29.35 [23.53 to 36.61] | 25.32 [18.6 to 34.47]

11. Secondary Outcome: Humoral Immune Response in Terms of Neutralising Antibodies Against the Flu A/Netherlands/602/2009 (H1N1) Vaccine Strain
Description: Antibody titers were expressed as Geometric mean titers (GMTs).
Time Frame: At Day 0, Day 21, Day 42 and Month 6
Population: The ATP cohort for immunogenicity including all evaluable subjects for whom assay results were available at the considered time points. No blood samples were taken at Day 0 and Day 21 and hence no GMTs computed for the Flu BS2 Groups. This analysis was conducted on a randomly selected subset of one third of the subjects.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 16 | 15 | 14 | 12 | 13 | 15
Titers
  H1N1, Day 0: number analyzed (Participants) | 16 | 15 | 14 | 0 | 0 | 0
  H1N1, Day 0 | 4.9 [3.9 to 6.1] | 7.1 [3.9 to 12.7] | 8 [3 to 21.3] |  |  |
  H1N1, Day 21: number analyzed (Participants) | 16 | 15 | 14 | 0 | 0 | 0
  H1N1, Day 21 | 27.7 [13 to 58.8] | 65.9 [24.6 to 176.4] | 109.4 [34.5 to 346.7] |  |  |
  H1N1, Day 42 | 433.2 [295.2 to 635.6] | 473.7 [301.5 to 744.1] | 438.4 [191.3 to 1004.8] | 533.4 [298.4 to 953.7] | 260.1 [141.9 to 476.6] | 199.5 [112.7 to 353.2]
  H1N1, Month 6 | 158.9 [110.4 to 228.8] | 203.3 [133.7 to 309.3] | 232.1 [81.8 to 658.4] | 156.6 [89.8 to 273.3] | 166 [88.7 to 310.6] | 150.9 [62.7 to 363.1]

12. Secondary Outcome: Humoral Immune Response in Terms of Neutralising Antibodies Against the Flu A/Netherlands/602/2009 (H1N1) Vaccine Strain
Description: Antibody titers were expressed as Geometric mean titers (GMTs).
Time Frame: At Month 12
Population: The ATP cohort for immunogenicity including all evaluable subjects for whom assay results were available at Month 12. No blood samples were planned at Month 12 the Flu BS1 Groups and hence no GMTs computed for these Groups. This analysis was conducted on a randomly selected subset of one third of the subjects.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 11 | 12 | 12
Titers | 152.3 [88.8 to 261] | 129.9 [71.2 to 236.8] | 138.3 [71.6 to 267.2]

13. Secondary Outcome: Number of Seroconverted Subjects for Neutralising Antibodies Against the Flu A/Netherlands/602/2009 (H1N1) Virus Strain
Description: as for outcome 2
Time Frame: At Day 21 and Day 42
Population: The ATP cohort for immunogenicity including subjects with assay results available for Day 0, Day 21 and Day 42. As no pre-vaccination (Day 0 and Day 21) blood samples were planned for the Flu BS2 Groups, seroconversion could not be computed for those groups. This analysis was conducted on a randomly selected subset of one third of the subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group
Number analyzed (Participants) | 16 | 15 | 14
Participants
  H1N1, Day 21 | 8 | 10 | 9
  H1N1, Day 42 | 15 | 15 | 14

14. Secondary Outcome: Number of Seroconverted Subjects for Neutralising Antibodies Against the Flu A/Netherlands/602/2009 (H1N1) Virus Strain
Description: as for outcome 2
Time Frame: At Month 6
Population: The ATP cohort for antibody persistence at Month 6 including subjects with assay results available for Day 0, Day 21 and Month 6. As no pre-vaccination (Day 0/21) blood samples were planned for the Flu BS2 Groups, seroconversion could not be computed for those groups. This analysis was done on a randomly selected subset of a third of the subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group
Number analyzed (Participants) | 16 | 15 | 13
Participants | 16 | 14 | 12

15. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as significant pain at rest that prevented normal everyday activities as assessed by inability to attend/do work or school or cried when limb was moved/spontaneously painful. Grade 3 redness and swelling was greater than 50 millimeters (mm) i.e. > 50mm.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The Total Vaccinated cohort including all vaccinated subjects who returned their symptom sheet.
Measure: Count of Participants; unit: Participants
Groups:
- Flu pooled_3-5 Years Group: Pooled data of subjects aged 3 to 5 years from the Flu BS1 and Flu BS2 Groups
- Flu pooled_6-9 Years Group: Pooled data of subjects aged 6 to 9 years from the Flu BS1 and Flu BS2 Groups
- Flu pooled_10-17 Years Group: Pooled data of subjects aged 10 to 17 years from the Flu BS1 and Flu BS2 Groups
Arm/Group | Flu pooled_3-5 Years Group | Flu pooled_6-9 Years Group | Flu pooled_10-17 Years Group
Number analyzed (Participants) | 60 | 65 | 118
Participants
  Any Pain | 40 | 49 | 96
  Grade 3 Pain | 4 | 9 | 11
  Any Redness | 28 | 28 | 46
  Grade 3 Redness | 4 | 2 | 4
  Any Swelling | 22 | 22 | 46
  Grade 3 Swelling | 2 | 3 | 10

16. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were arthralgia, diarrhoea, drowsiness, fatigue, gastro-intestinal symptoms, headache, irritability, loss of appetite, myalgia, shivering, sweating and fever [axillary temperature above 37.5 degrees Celsius (°C)]. Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature above 39.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The Total Vaccinated cohort including all vaccinated subjects who returned their symptom sheet.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu pooled_3-5 Years Group | Flu pooled_6-9 Years Group | Flu pooled_10-17 Years Group
Number analyzed (Participants) | 60 | 65 | 118
Participants
  Any Arthralgia | 0 | 14 | 25
  Grade 3 Arthralgia | 0 | 1 | 3
  Related Arthralgia | 0 | 14 | 23
  Any Diarrhoea | 9 | 0 | 0
  Grade 3 Diarrhoea | 2 | 0 | 0
  Related Diarrhoea | 5 | 0 | 0
  Any Drowsiness | 20 | 0 | 0
  Grade 3 Drowsiness | 3 | 0 | 0
  Related Drowsiness | 18 | 0 | 0
  Any Fatigue | 0 | 24 | 53
  Grade 3 Fatigue | 0 | 4 | 6
  Related Fatigue | 0 | 23 | 50
  Any Gastro-intestinal symptoms | 0 | 13 | 30
  Grade 3 Gastro-intestinal symptoms | 0 | 1 | 5
  Related Gastro-intestinal symptoms | 0 | 10 | 23
  Any Headache | 0 | 19 | 61
  Grade 3 Headache | 0 | 4 | 10
  Related Headache | 0 | 19 | 56
  Any Irritability | 18 | 0 | 0
  Grade 3 Irritability | 1 | 0 | 0
  Related Irritability | 18 | 0 | 0
  Any Loss of appetite | 18 | 0 | 0
  Grade 3 Loss of appetite | 1 | 0 | 0
  Related Loss of appetite | 17 | 0 | 0
  Any Myalgia | 0 | 13 | 45
  Grade 3 Myalgia | 0 | 1 | 3
  Related Myalgia | 0 | 13 | 43
  Any Shivering | 10 | 10 | 35
  Grade 3 Shivering | 0 | 0 | 3
  Related Shivering | 9 | 9 | 33
  Any Sweating | 9 | 10 | 18
  Grade 3 Sweating | 0 | 0 | 1
  Related Sweating | 8 | 9 | 15
  Any Fever (≥37.5°C) | 27 | 13 | 30
  Grade 3 Fever (>39°C) | 4 | 3 | 4
  Related Fever | 23 | 11 | 23

17. Secondary Outcome: Number of Subjects Reporting Any Medically Attended Adverse Events (MAEs)
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination.
Time Frame: During the entire study period (Day 0 to Month 12)
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 31 | 31 | 60 | 30 | 34 | 58
Participants | 22 | 19 | 36 | 24 | 16 | 34

18. Secondary Outcome: Number of Subjects Reporting Any Adverse Events of Specific Interest (AESI)/Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) were defined as a subset of adverse events that included both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which might or might not have an autoimmune etiology. "Any pIMD" was defined as at least one pIMD experienced by the study subject.
Time Frame: During the entire study period (Day 0 to Month 12)
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu pooled_3-5 Years Group | Flu pooled_6-9 Years Group | Flu pooled_10-17 Years Group
Number analyzed (Participants) | 61 | 65 | 118
Participants | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: Within the 84-day after the first vaccination or from 63-day follow-up period after the second vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu pooled_3-5 Years Group | Flu pooled_6-9 Years Group | Flu pooled_10-17 Years Group
Number analyzed (Participants) | 61 | 65 | 118
Participants
  Any AE(s) | 42 | 25 | 53
  Grade 3 AE(s) | 3 | 1 | 5
  Related AE(s) | 9 | 2 | 4

20. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 to Month 12)
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 31 | 31 | 60 | 30 | 34 | 58
Participants
  Any SAE(s) | 1 | 1 | 1 | 1 | 0 | 3
  Related SAE(s) | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects With Normal and Abnormal Haematological and Biochemistry Parameters With Respect to Alanine Aminotransferase (ALAT), Aspartate Aminotransferase (ASAT), Total Bilirubin, Bilirubin Conjugated/ Direct,Creatine and Blood Urea Nitrogen(BUN)
Description: Subjects were categorized by age and according to their results at pre-vaccination (Day 0), Day 21, Day 42 and Month 6 which were below, within and above the normal ranges or unknown as measured by validated assay according to international standards.
Time Frame: At Day 0, Day 21, Day 42 and Month 6 (M6)
Population: The Total Vaccinated cohort including all vaccinated subjects with data available for the respective assays at the considered timepoints. Note that for Flu BS2 Groups, no blood samples were taken at Day 0 and Day 21 and hence no data for these timepoints are reported for the Flu BS2 Groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Number analyzed (Participants) | 31 | 31 | 60 | 26 | 33 | 58
Participants
  ALAT, Day 0 Unknown: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  ALAT, Day 0 Unknown | 1 | 1 | 1 |  |  |
  ALAT, Day 0 Below: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  ALAT, Day 0 Below | 0 | 0 | 0 |  |  |
  ALAT, Day 0 Within: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  ALAT, Day 0 Within | 29 | 30 | 58 |  |  |
  ALAT, Day 0 Above: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  ALAT, Day 0 Above | 0 | 0 | 1 |  |  |
  ALAT, Day 21 Unknown: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  ALAT, Day 21 Unknown | 1 | 0 | 1 |  |  |
  ALAT, Day 21 Below: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  ALAT, Day 21 Below | 0 | 0 | 0 |  |  |
  ALAT, Day 21 Within: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  ALAT, Day 21 Within | 30 | 30 | 58 |  |  |
  ALAT, Day 21 Above: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  ALAT, Day 21 Above | 0 | 0 | 0 |  |  |
  ALAT, Day 42 Unknown: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  ALAT, Day 42 Unknown | 0 | 0 | 2 | 0 | 0 | 0
  ALAT, Day 42 Below: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  ALAT, Day 42 Below | 0 | 0 | 0 | 0 | 0 | 0
  ALAT, Day 42 Within: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  ALAT, Day 42 Within | 31 | 30 | 55 | 26 | 32 | 56
  ALAT, Day 42 Above: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  ALAT, Day 42 Above | 0 | 0 | 1 | 0 | 1 | 1
  ALAT, M6 Unknown: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  ALAT, M6 Unknown | 0 | 0 | 1 | 0 | 0 | 0
  ALAT, M6 Below: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  ALAT, M6 Below | 0 | 0 | 0 | 0 | 0 | 0
  ALAT, M6 Within: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  ALAT, M6 Within | 30 | 29 | 56 | 24 | 29 | 52
  ALAT, M6 Above: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  ALAT, M6 Above | 0 | 0 | 1 | 0 | 0 | 1
  ASAT, Day 0 Unknown: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  ASAT, Day 0 Unknown | 1 | 1 | 1 |  |  |
  ASAT, Day 0 Below: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  ASAT, Day 0 Below | 0 | 0 | 0 |  |  |
  ASAT, Day 0 Within: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  ASAT, Day 0 Within | 26 | 29 | 58 |  |  |
  ASAT, Day 0 Above: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  ASAT, Day 0 Above | 3 | 1 | 1 |  |  |
  ASAT, Day 21 Unknown: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  ASAT, Day 21 Unknown | 1 | 0 | 1 |  |  |
  ASAT, Day 21 Below: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  ASAT, Day 21 Below | 0 | 0 | 0 |  |  |
  ASAT, Day 21 Within: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  ASAT, Day 21 Within | 30 | 29 | 58 |  |  |
  ASAT, Day 21 Above: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  ASAT, Day 21 Above | 0 | 1 | 0 |  |  |
  ASAT, Day 42 Unknown: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  ASAT, Day 42 Unknown | 0 | 1 | 2 | 0 | 0 | 0
  ASAT, Day 42 Below: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  ASAT, Day 42 Below | 0 | 0 | 0 | 0 | 0 | 0
  ASAT, Day 42 Within: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  ASAT, Day 42 Within | 31 | 29 | 55 | 25 | 31 | 55
  ASAT, Day 42 Above: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  ASAT, Day 42 Above | 0 | 0 | 1 | 1 | 2 | 2
  ASAT, M6 Unknown: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  ASAT, M6 Unknown | 0 | 0 | 1 | 0 | 0 | 0
  ASAT, M6 Below: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  ASAT, M6 Below | 0 | 0 | 0 | 0 | 0 | 0
  ASAT, M6 Within: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  ASAT, M6 Within | 30 | 28 | 57 | 24 | 29 | 50
  ASAT, M6 Above: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  ASAT, M6 Above | 0 | 1 | 0 | 0 | 0 | 3
  Total Bilirubin, Day 0 Unknown: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Total Bilirubin, Day 0 Unknown | 1 | 1 | 1 |  |  |
  Total Bilirubin, Day 0 Below: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Total Bilirubin, Day 0 Below | 0 | 0 | 0 |  |  |
  Total Bilirubin, Day 0 Within: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Total Bilirubin, Day 0 Within | 29 | 28 | 57 |  |  |
  Total Bilirubin, Day 0 Above: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Total Bilirubin, Day 0 Above | 0 | 2 | 2 |  |  |
  Total Bilirubin, Day 21 Unknown: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Total Bilirubin, Day 21 Unknown | 1 | 0 | 1 |  |  |
  Total Bilirubin, Day 21 Below: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Total Bilirubin, Day 21 Below | 0 | 0 | 0 |  |  |
  Total Bilirubin, Day 21 Within: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Total Bilirubin, Day 21 Within | 30 | 28 | 55 |  |  |
  Total Bilirubin, Day 21 Above: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Total Bilirubin, Day 21 Above | 0 | 2 | 3 |  |  |
  Total Bilirubin, Day 42 Unknown: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Total Bilirubin, Day 42 Unknown | 0 | 0 | 2 | 0 | 0 | 0
  Total Bilirubin, Day 42 Below: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Total Bilirubin, Day 42 Below | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Day 42 Within: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Total Bilirubin, Day 42 Within | 31 | 30 | 55 | 26 | 33 | 55
  Total Bilirubin, Day 42 Above: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Total Bilirubin, Day 42 Above | 0 | 0 | 1 | 0 | 0 | 2
  Total Bilirubin, M6 Unknown: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Total Bilirubin, M6 Unknown | 0 | 0 | 1 | 0 | 0 | 0
  Total Bilirubin, M6 Below: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Total Bilirubin, M6 Below | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, M6 Within: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Total Bilirubin, M6 Within | 30 | 28 | 55 | 24 | 29 | 51
  Total Bilirubin, M6 Above: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Total Bilirubin, M6 Above | 0 | 1 | 2 | 0 | 0 | 2
  Bilirubin Conjugated / Direct, Day 0 Unknown: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 0 Unknown | 1 | 1 | 1 |  |  |
  Bilirubin Conjugated / Direct, Day 0 Below: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 0 Below | 0 | 0 | 0 |  |  |
  Bilirubin Conjugated / Direct, Day 0 Within: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 0 Within | 29 | 30 | 58 |  |  |
  Bilirubin Conjugated / Direct, Day 0 Above: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 0 Above | 0 | 0 | 1 |  |  |
  Bilirubin Conjugated / Direct, Day 21 Unknown: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 21 Unknown | 1 | 0 | 1 |  |  |
  Bilirubin Conjugated / Direct, Day 21 Below: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 21 Below | 0 | 0 | 0 |  |  |
  Bilirubin Conjugated / Direct, Day 21 Within: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 21 Within | 30 | 30 | 58 |  |  |
  Bilirubin Conjugated / Direct, Day 21 Above: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 21 Above | 0 | 0 | 0 |  |  |
  Bilirubin Conjugated / Direct, Day 42 Unknown: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Bilirubin Conjugated / Direct, Day 42 Unknown | 0 | 0 | 2 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 42 Below: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Bilirubin Conjugated / Direct, Day 42 Below | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, Day 42 Within: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Bilirubin Conjugated / Direct, Day 42 Within | 31 | 30 | 56 | 26 | 33 | 57
  Bilirubin Conjugated / Direct, Day 42 Above: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Bilirubin Conjugated / Direct, Day 42 Above | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, M6 Unknown: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Bilirubin Conjugated / Direct, M6 Unknown | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, M6 Below: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Bilirubin Conjugated / Direct, M6 Below | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin Conjugated / Direct, M6 Within: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Bilirubin Conjugated / Direct, M6 Within | 30 | 29 | 57 | 24 | 29 | 53
  Bilirubin Conjugated / Direct, M6 Above: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Bilirubin Conjugated / Direct, M6 Above | 0 | 0 | 0 | 0 | 0 | 0
  Creatine, Day 0 Unknown: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Creatine, Day 0 Unknown | 1 | 1 | 1 |  |  |
  Creatine, Day 0 Below: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Creatine, Day 0 Below | 2 | 0 | 1 |  |  |
  Creatine, Day 0 Within: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Creatine, Day 0 Within | 27 | 29 | 52 |  |  |
  Creatine, Day 0 Above: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  Creatine, Day 0 Above | 0 | 1 | 6 |  |  |
  Creatine, Day 21 Unknown: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Creatine, Day 21 Unknown | 1 | 0 | 1 |  |  |
  Creatine, Day 21 Below: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Creatine, Day 21 Below | 3 | 0 | 4 |  |  |
  Creatine, Day 21 Within: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Creatine, Day 21 Within | 27 | 28 | 48 |  |  |
  Creatine, Day 21 Above: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  Creatine, Day 21 Above | 0 | 2 | 6 |  |  |
  Creatine, Day 42 Unknown: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Creatine, Day 42 Unknown | 0 | 0 | 2 | 0 | 0 | 0
  Creatine, Day 42 Below: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Creatine, Day 42 Below | 2 | 1 | 3 | 0 | 1 | 2
  Creatine, Day 42 Within: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Creatine, Day 42 Within | 28 | 29 | 52 | 24 | 31 | 51
  Creatine, Day 42 Above: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  Creatine, Day 42 Above | 1 | 0 | 1 | 2 | 1 | 4
  Creatine, M6 Unknown: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Creatine, M6 Unknown | 0 | 0 | 1 | 0 | 0 | 0
  Creatine, M6 Below: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Creatine, M6 Below | 1 | 1 | 2 | 1 | 0 | 5
  Creatine, M6 Within: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Creatine, M6 Within | 28 | 28 | 55 | 22 | 29 | 47
  Creatine, M6 Above: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  Creatine, M6 Above | 1 | 0 | 0 | 1 | 0 | 1
  BUN, Day 0 Unknown: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  BUN, Day 0 Unknown | 1 | 1 | 1 |  |  |
  BUN, Day 0 Below: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  BUN, Day 0 Below | 0 | 0 | 2 |  |  |
  BUN, Day 0 Within: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  BUN, Day 0 Within | 28 | 30 | 57 |  |  |
  BUN, Day 0 Above: number analyzed (Participants) | 30 | 31 | 60 | 0 | 0 | 0
  BUN, Day 0 Above | 1 | 0 | 0 |  |  |
  BUN, Day 21 Unknown: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  BUN, Day 21 Unknown | 1 | 0 | 1 |  |  |
  BUN, Day 21 Below: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  BUN, Day 21 Below | 1 | 2 | 3 |  |  |
  BUN, Day 21 Within: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  BUN, Day 21 Within | 29 | 27 | 55 |  |  |
  BUN, Day 21 Above: number analyzed (Participants) | 31 | 30 | 59 | 0 | 0 | 0
  BUN, Day 21 Above | 0 | 1 | 0 |  |  |
  BUN, Day 42 Unknown: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  BUN, Day 42 Unknown | 0 | 0 | 2 | 0 | 0 | 0
  BUN, Day 42 Below: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  BUN, Day 42 Below | 1 | 2 | 1 | 1 | 0 | 0
  BUN, Day 42 Within: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  BUN, Day 42 Within | 29 | 28 | 55 | 23 | 32 | 56
  BUN, Day 42 Above: number analyzed (Participants) | 31 | 30 | 58 | 26 | 33 | 57
  BUN, Day 42 Above | 1 | 0 | 0 | 2 | 1 | 1
  BUN, M6 Unknown: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  BUN, M6 Unknown | 1 | 0 | 1 | 0 | 0 | 0
  BUN, M6 Below: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  BUN, M6 Below | 1 | 0 | 2 | 0 | 0 | 0
  BUN, M6 Within: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  BUN, M6 Within | 27 | 28 | 54 | 24 | 27 | 53
  BUN, M6 Above: number analyzed (Participants) | 30 | 29 | 58 | 24 | 29 | 53
  BUN, M6 Above | 1 | 1 | 1 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: SAEs:During the entire study period (Day 0 to Month 6), Solicited local and general symptoms:During the 7-day (Days 0-6) post-vaccination period;Unsolicited symptoms:Within the 84-day or from 63-day follow-up period after the 1st and 2nd dose,respectively.
Arm/Group | Flu BS1_3-5 Years Group | Flu BS1_6-9 Years Group | Flu BS1_10-17 Years Group | Flu BS2_3-5 Years Group | Flu BS2_6-9 Years Group | Flu BS2_10-17 Years Group
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/31 | 1/60 | 1/30 | 0/34 | 3/58
Other Adverse Events (participants affected / at risk) | 30/31 | 25/31 | 56/60 | 26/30 | 26/34 | 50/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flu BS1_3-5 Years Group (N=31) | Flu BS1_6-9 Years Group (N=31) | Flu BS1_10-17 Years Group (N=60) | Flu BS2_3-5 Years Group (N=30) | Flu BS2_6-9 Years Group (N=34) | Flu BS2_10-17 Years Group (N=58)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ranula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flu BS1_3-5 Years Group (N=31) | Flu BS1_6-9 Years Group (N=31) | Flu BS1_10-17 Years Group (N=60) | Flu BS2_3-5 Years Group (N=30) | Flu BS2_6-9 Years Group (N=34) | Flu BS2_10-17 Years Group (N=58)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (10) | 11 (14) | 2 (2) | 7 (9) | 14 (17)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Chills (General disorders) | 7 (11) | 7 (8) | 18 (24) | 3 (4) | 3 (4) | 17 (22)
Conjunctivitis (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (1) | 0 (0) | 5 (10) | 2 (3) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 10 (12) | 0 (0) | 1 (1) | 9 (13) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 14 (18) | 16 (20) | 23 (34) | 14 (21) | 12 (16) | 23 (30)
Fatigue (General disorders) | 0 (0) | 13 (18) | 29 (37) | 0 (0) | 11 (15) | 24 (36)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 7 (11) | 18 (21) | 0 (0) | 6 (7) | 12 (13)
Headache (Nervous system disorders) | 1 (1) | 9 (14) | 30 (47) | 4 (4) | 10 (13) | 31 (50)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 9 (10) | 5 (6) | 6 (6) | 9 (10)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Irritability (Psychiatric disorders) | 9 (13) | 0 (0) | 0 (0) | 9 (14) | 0 (0) | 0 (0)
Lice infestation (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (10) | 21 (26) | 1 (1) | 7 (12) | 24 (29)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 3 (4) | 4 (6) | 2 (2) | 4 (5)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 19 (29) | 24 (40) | 51 (92) | 21 (38) | 25 (42) | 45 (75)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 15 (22) | 7 (10) | 19 (22) | 15 (22) | 9 (11) | 12 (14)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 11 (16) | 0 (0) | 0 (0) | 9 (11) | 0 (0) | 0 (0)
Swelling (General disorders) | 13 (16) | 13 (18) | 21 (28) | 9 (13) | 9 (13) | 25 (38)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (2) | 5 (5) | 4 (5) | 0 (0) | 2 (3)
Viral infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.